CLINICAL TRIAL: NCT07081178
Title: A Non-interventional Study Investigating Semaglutide in Combination With Lifestyle-based Modifications for the Management of Obesity in Real-World Clinical Practice in Germany Non-interventional.
Brief Title: A Non-interventional Study Investigating Semaglutide in Combination With Lifestyle-based Modifications for the Management of Obesity in Real-World Clinical Practice in Germany (WeGo Real Germany).
Acronym: WeGoReal
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-8332; U1111-1314-8335 (Other: WHO)
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants will be treated with commercially available semaglutide along with lifestyle modification in the routine clinical practice.
  Interventions: Drug: Semaglutide
- Group B: Participants with lifestyle modification in the routine clinical practice will be included.

INTERVENTIONS:
Drug: Semaglutide — Semaglutide injection will be self-administered once weekly subcutaneously at any time of the day with or without meals.
  Groups: Group A

SUMMARY:
Participants will be treated with commercially available semaglutide according to routine clinical practice at the discretion of the treating physician for the management of obesity. The purpose of this study is to collect data on the effect of Semaglutide under everyday conditions in participants. Participants and doctor had already decided that they will get semaglutide prescribed by doctor, independently of patient's participation in this study. The study will last for 12 months.

ELIGIBILITY:
Common inclusion criteria for Group A and Group B:

1. Male or female, age above or equal to 18 years at the time signing informed consent.
2. Body mass index (BMI) more than or equal to (≥) 30 kilogram per meter square (kg/m^2) with at least one of the following diagnosed obesity-related comorbidities:

   arterial hypertension, pre-diabetes, Obstructive Sleep Apnea (OSA) or coronary heart disease, chronic heart failure, or BMI ≥35 kg/m^2.
3. History of at least one self-reported unsuccessful attempt to lose weight.
4. Capable of completing informed consent.

Additional inclusion criteria for Group A:

1. The decision to initiate treatment with commercially available Wegovy has been made by the participant and the treating physician before and independently from the decision to include the participant in this study.
2. Initiation of treatment is not modified in any case due to participant's participation in the study.

Common exclusion criteria for Group A and Group B:

1. Previous participation in this study (participation is defined as having given informed consent in this study)
2. Treatment with an investigational drug within 30 days prior to enrolment into the study.
3. Participant has had a prior serious allergic reaction to semaglutide or any of the ingredients in Wegovy.
4. Women with pregnancy or breast-feeding.
5. Women of childbearing potential and not using an adequate contraceptive method.
6. Men and women in their pregnancy attempts.
7. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
8. History of any Glucagon-like peptide-1 (GLP-1) treatment within 180 days.
9. History of type 1 or type 2 diabetes mellitus.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two groups of participants are planned to be included, one Group (A) with those initiating semaglutide adjunct with lifestyle modification, and the other Group (B) with those only with lifestyle modification.
Sampling Method: Non-Probability Sample
Enrollment: 555 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-10-21 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
Change in relative body weight | From baseline to month 6 and month 9
  Percentage (%)

SECONDARY OUTCOMES:
Change in relative body weight | From baseline to month 3 and 12
  Percentage (%)
Change in body weight | from baseline to month 3, month 6, month 9 and month 12
  Kilogram (Kg)
Change in Haemoglobin A1c (HbA1c) | from baseline to month 3, month 6, month 9 and month 12
  millimoles per mole (mmol/mol)
Change in fasting plasma glucose (FPG) | from baseline to month 3, month 6, month 9 and month 12
  milligram per deciliter (mg/dL)
Change in total cholesterol | from baseline to month 3, month 6, month 9 and month 12
  mg/dL
Change in high density lipoprotein (HDL) | from baseline to month 3, month 6, month 9 and month 12
  mg/dL
Change in low density lipoprotein (LDL) | from baseline to month 3, month 6, month 9 and month 12
  mg/dL
Change in very low density lipoprotein (VLDL) | from baseline to month 3, month 6, month 9 and month 12
  mg/dL
Change in lipoprotein A [Lp(a)] | from baseline to month 3, month 6, month 9 and month 12
  mg/dL
Change in triglycerides | from baseline to month 3, month 6, month 9 and month 12
  mg/dL
Change in estimated glomerular filtration rate (eGFR) eGFR | from baseline to month 3, month 6, month 9 and month 12
  milliliters per minute per 1.73 square meters (mL/min/1.73m²)
Change in waist circumference | from baseline to month 3, month 6, month 9 and month 12
  Centimeter (cm)
Change in systolic blood pressure (SBP) | from baseline to month 3, month 6, month 9 and month 12
  millimeters of mercury (mmHg)
Change in diastolic blood pressure (DBP) | from baseline to month 3, month 6, month 9 and month 12
  mmHg
Change in C-reactive protein (CRP) or high-sensitivity C-reactive protein (hs-CRP) | from baseline to month 3, month 6, month 9 and month 12
  milligrams per liter (mg/L)
Change in platelet count | from baseline to month 3, month 6, month 9 and month 12
  number of platelets per liter (10^9/L)
Change in gamma-glutamyl transferase (GGT) | from baseline to month 3, month 6, month 9 and month 12
  unit per liter (U/L)
Change in alanine aminotransferase/serum glutamic-pyruvic transaminase (ALT/GPT) | from baseline to month 3, month 6, month 9 and month 12
  units per liter (U/L)
Change in aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/GOT) | from baseline to month 3, month 6, month 9 and month 12
  units per liter (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com